CLINICAL TRIAL: NCT06327724
Title: The Effects of Belimumab on Synovial Inflammation and Composition of Lymph Nodes in SLE Patients
Brief Title: Belimumab in SLE Synovial Inflammation and Lymph Nodes
Status: Recruiting | Type: Observational
Sponsor: Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA) (Other)
Collaborators: GlaxoSmithKline (Industry)
Responsible Party: Principal Investigator, Sander Tas, Prof. dr., Academisch Medisch Centrum - Universiteit van Amsterdam (AMC-UvA)
Other Study IDs: 12434
Record Dates: First submitted 2024-03-13; First posted 2024-03-25 (Actual); Last update posted 2024-03-25 (Actual); Status verified 2024-03

CONDITIONS: Systemic Lupus Erythematosus
Keywords: lymph node; synovial tissue
MeSH Terms: conditions — Lupus Erythematosus, Systemic | interventions — belimumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — PBMC Lymph node biopsy Synovial tissue biopsy
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

INTERVENTIONS:
Drug: Belimumab — Start of new treatment due to active disease
  Other Names: Any other treatment

SUMMARY:
Systemic lupus erythematosus (SLE)is an immune-mediated inflammatory disease (IMIDs) of which the cellular and molecular alterations of the immune system driving the diseases still remains largely unknown. Accordingly, it remains difficult to predict the individual patient's response to treatment. Moreover, the patient's response to treatment remains heterogeneous and difficult to predict, despite the development of a variety of novel and powerful drugs (including the so-called biologicals). Therefore, there is a clear need for the identification and validation of cellular and molecular biomarkers which can provide useful clinical information for diagnosis, classification, prognosis and treatment, as well as the development of new therapeutic strategies. Biomarkers can be found and analyzed in different body compartments, of which the peripheral blood and the intra-articular synovial fluid or tissue are most easily accessible. However, previous studies in RA and other IMIDs showed that adaptive immune responses in other tissues such as lymph nodes also play an important role. Investigating other immune compartments of the body such as the lymph nodes could result in new insights. To study the early pathogenesis of inflammatory conditions, in 2008 our department initiated core-needle inguinal lymph node biopsy sampling. Since then more than 100 lymph node biopsy procedures were performed. The procedure is well-tolerated and, other than a small hematoma which does not require therapy in most of the cases, no complications were reported.

In the current study, the effects of belimumab (anti-BAFF) in SLE will be investigated by studying the immune alterations taking place in lymph nodes in comparison to peripheral blood and immune alterations taking place in the end-organ, e.g. the joint (wrist, knee or ankle) by taking synovial biopsies during a needle- or mini-arthroscopy. This procedure has been performed frequently in our department over the last 15 years. In this way immune alterations in the lymph nodes (secondary lymphoid organ), peripheral blood (systemic) and the joint (end organ for the disease) will be assessed and compared.

DETAILED DESCRIPTION:
The primary goal of this study is to investigate the effects of belimumab on the composition of lymph nodes and the inflamed synovial tissue as well as (subsets of) immune cells in the peripheral blood using advanced flow cytometry methods. In addition, immunological alterations in lymphoid tissue and inflamed synovial tissue of SLE patients will be identified and correlated with disease stage/phenotype, prognosis, and belimumab treatment response. In this way novel biomarkers may be identified and validated that can be used for personalized medicine in SLE.

The specific types of immunological alterations that will be studied include:

* Genetic, epigenetic and transcriptional alterations of immune cells and stromal cells, including single cell RNA sequencing (scRNAseq)
* TCR and BCR repertoire
* Phenotype and function of (auto-reactive) T and B cells
* Cytokine production by immune cells and stromal cells
* Signalling events in immune cells and stromal cells
* Antigen presentation by immune cells and stromal cells

All of these parameters will be compared between lymph nodes, blood and synovium (if applicable) in SLE patients before and after belimumab treatment.

Research Hypothesis Patients with SLE contain activated immune cells in their lymph nodes and inflamed synovial tissue. Furthermore, activation of stromal cells such as fibroblasts and endothelial cells may also be increased compared to (historical) healthy controls. In addition, dominant T cell and B cell clones may be present. Belimumab treatment will result in reduced inflammation in the synovial tissue and perhaps even normalization of lymph node architecture.

ELIGIBILITY:
Inclusion Criteria:

SLE patients who:

1. fulfill ACR 1997 and/or SLICC and/or ACR/ EULAR 2019 criteria,
2. have active joint disease (arthritis) in wrist, knee or ankle joints.
3. have a SLEDAI-2K score ≥6.
4. are aged between 18-75
5. start with belimumab or any other immunosuppressive treatment

Exclusion Criteria:

* Patients who are not able to give informed consent.
* Pregnancy
* Severe renal impairment (eGFR <30ml/min/1.73m2)
* Active nephritis
* Present or previous treatment with any cell depleting therapies, including anti-B-cell therapy or other investigational agents
* Intravenous cyclophosphamide 90 days prior to belimumab
* Any non-biologic investigational agent 30 Days Prior to belimumab (or 5 half-lives, whichever is greater)
* Live vaccines within 30 days prior to baseline or concurrently with belimumab
* Presence of any other disease for which study subjects need chronic or intermittent immunosuppressive therapy (e.g. prednisolon for COPD).
* History of malignancies neoplasm within the last 5 years except basal cell or squamous cell carcinoma of the skin treated with local resection only or carcinoma in situ of the uterine cervix treated locally and with no evidence of metastatic disease for 3 years
* Have any intercurrent significant medical or psychiatric illness that the investigator considers would make the candidate unsuitable for the study, including evidence of serious suicide risk including any history of suicidal behaviour in the last 6 months and/or any suicidal ideation in the last 2 months or who in the investigator's judgment, poses a significant suicide risk
* Have current drug or alcohol abuse or dependence, or a history of drug or alcohol abuse or dependence within 365 days prior to Day 0
* Have a historically positive HIV test or test positive at screening for HIV, or other immunodeficiency

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: SLE patients
Sampling Method: Non-Probability Sample
Enrollment: 15 (Estimated)
Dates: Start 2023-09-01 (Actual); Primary Completion 2025-01-01 (Estimated); Study Completion 2025-03-01 (Estimated)

PRIMARY OUTCOMES:
Differences in lymph node cellular composition as assessed by advanced flow cytometry | 4 weeks
  Differences in lymph node cellular composition and functional aspects in SLE patients after belimumab treatment compared to SLE patients starting any other effective treatment.

SECONDARY OUTCOMES:
Differences in peripheral blood cellular composition as assessed by advanced flow cytometry | 4 weeks
  Differences in peripheral blood cellular composition and functional aspects in SLE patients after belimumab treatment compared to SLE patients starting any other effective treatment.
Differences in synovial tissue cellular composition as assessed by advanced flow cytometry | 4 weeks
  Differences in synovial tissue cellular composition and functional aspects in SLE patients after belimumab treatment compared to SLE patients starting any other effective treatment.

CONTACTS AND LOCATIONS:
Locations (1):
- Amsterdam UMC; location Academic Medical Center, Amsterdam, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided